CLINICAL TRIAL: NCT06490978
Title: Predictors of Early Hematoma Expansion in Patients With Acute Intracerebral Hemorrhage (Clinical and Laboratory Study)
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hussein Abd El-samee, Resident doctor, Assiut University
Other Study IDs: ICH Expansion
Record Dates: First submitted 2024-02-27; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: ICH - Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: CT Brain — Patient needs follow up ct brain , cbc , CRP

SUMMARY:
This study aim to develop inflammatory score based on proper integration of several inflammatory markers and investigate whether it was associated with hematoma expansion and poor outcomes in patients with ICH .

DETAILED DESCRIPTION:
Intracerebral hemorrhage(ICH) accounts for approximately a quarter of all stroke subtypes with high mortality and the survi- vors always have varying degrees of residual disability. However, few medical and surgical treatments are clearly beneficial comparing with ischemic stroke. Hematoma expansion, which is a determinant of poor outcomes, occurs in about 30% of ICH patients especially at the early stage. Attenuating hema- toma expansion is a compelling target for ICH treatment, while the outcomes have not been accordingly improved after curbing the growth of hematoma in several clinical trials. It will be more helpful if a predictor can identify the risk of hematoma expansion and poor outcome rapidly and accurately. Thus the antiexpansion treatment to the patients with positive of such predictor is likely to provide clinical benefits.

ELIGIBILITY:
Inclusion Criteria:

* patients having spontaneous ICH aged 18 years or older admitted to a stroke unit within 24 hours After symptom onset .

Exclusion Criteria:

1- patient have secondary ICH (cerebral aneurysm, Moyamoya syndrome, arteriovenous malformation, tumor, trauma or hemorrhagic transformation from brain infarction); (2)patient have primary intraventricular hemorrhage (IVH); (3)patients with historical modified Rankin scale (mRS) score greater than 1 (4) patient refused to be enrolled.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Spontaneous ICH patients aged 18 years or older admitted to a stroke unit within 24 hours After symptom onset .approximately a quarter of all stroke subtypes with high mortality and the survi- vors always have varying degrees of residual disability. However, few medical and surgical treatments are clearly beneficial comparing with ischemic stroke. Hematoma expansion, which is a determinant of poor outcomes, occurs in about 30% of ICH patients especially at the early stage. Attenuating hema- toma expansion is a compelling target for ICH treatment, while the outcomes have not been accordingly improved after curbing the growth of hematoma in several clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
primary (main): appropriate predictor of hematoma expansion and poor outcomes with good accuracies. | Baseline
  The current study suggests inflammatory score consisting of appropriate integration of NLR, PLR, MLR, SII, LDH, and CRP is independently associated with hematoma expansion and poor outcomes of different terms in ICH patients, including secondary neurological deterioration within 48 hours, 30-day mortality, and 3-month poor mRS. Moreover, inflammatory score greater than or equal to 5 is validated as an appropriate predictor of hematoma expansion and poor outcomes with good accuracies

SECONDARY OUTCOMES:
Secondary outcome | One year
  Secondary (subsidiary) :
  1. inflammatory score based on proper integration of several inflammatory markers
  2. investigate whether it was associated with hematoma expansion in patients with ICH Helping . in better outcome and good prognosis
  3. prediction of secondary neurological deterioration within 48 hours, 30-day mortality, and 3- month poor mRS
  Secondary (subsidiary) :
  1. inflammatory score based on proper integration of several inflammatory markers
  2. investigate whether it was associated with hematoma expansion in patients with ICH Helping . in better outcome and good prognosis
  3. prediction of secondary neurological deterioration within 48 hours, 30-day mortality, and 3- month poor mRS

CONTACTS AND LOCATIONS:
Overall Officials: Amal M. Tohamy, Lecturer, Study Director — Assiut University; Ahmed M. Tawfik, Lecturer, Study Director — Assiut University